CLINICAL TRIAL: NCT07100444
Title: Spinal Metastasis as the First Presentation of Lung Malignancy: Clinical Characteristics and Postoperative Survival
Status: Completed | Type: Observational
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Yu Zhang, PhD, Professor, Guangdong Provincial People's Hospital
Other Study IDs: lungfirstboneMetas
Record Dates: First submitted 2025-07-24; First posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Lung Cancers; Bone Metastasis
Keywords: lung cancers; bone metastasis; spinal metastasis; postoperative survival outcomes
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Spinal Metastasis as the First Presentation of Lung Malignancy: It refers to patients who first present with symptoms such as pain or spinal cord compression caused by spinal metastasis, leading to the initial detection of bone metastasis, and are subsequently diagnosed with lung cancer.
- lung cancer who subsequently developed spinal metastasis: It refers to patients with a history of treatment for primary lung cancer who subsequently developed spinal metastasis during the course of the disease.

SUMMARY:
The aim of this study is to compare the clinical features and postoperative survival outcomes between patients with spinal metastasis as the initial manifestation of malignancy and those with spinal metastasis occurring after an established diagnosis of malignancy.

DETAILED DESCRIPTION:
The aim of this study is to compare the clinical features and postoperative survival outcomes between patients with spinal metastasis as the initial manifestation of malignancy and those with spinal metastasis occurring after an established diagnosis of malignancy. By analyzing and contrasting these two groups, we seek to identify any distinctive characteristics, prognostic factors, and potential implications for early detection and treatment strategies in patients with malignant spinal metastases.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Pathologically or radiologically confirmed diagnosis of lung cancer with spinal metastasis.
3. Patients with spinal metastasis who underwent surgical intervention.
4. Adequate medical records and follow-up data available.

Exclusion Criteria:

1. Patients with spinal metastasis originating from non-lung primary tumors.
2. Patients who did not receive surgical treatment for spinal metastasis.
3. Incomplete clinical data or lost to follow-up.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of adult patients diagnosed with lung cancer who have developed spinal metastasis. Participants will be selected from individuals treated at Guangdong Provincial People's Hospital. Eligible patients must have a diagnosis of lung cancer with spinal metastasis confirmed by pathological examination or imaging studies, and must have undergone surgical intervention for spinal metastasis.
Sampling Method: Non-Probability Sample
Enrollment: 139 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2025-03-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Postoperative Overall Survival | From the date of surgery until death or last follow-up, up to 5 years
  Postoperative overall survival is defined as the time from the date of surgery for spinal metastasis to the date of death from any cause. Patients who are still alive at the last follow-up will be censored at that date. Survival status will be ascertained by clinical follow-up and/or review of medical records.

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because of patient privacy concerns and local data protection regulations. Data may contain sensitive personal information that cannot be sufficiently anonymized to ensure participant confidentiality.